CLINICAL TRIAL: NCT03996720
Title: Integration of Metabolic and Inflammatory Mediator Profiles as a Potential Diagnostic Approach for Severe Sepsis in PICU
Brief Title: Early Identification and Effective Management of Pediatric Sepsis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Shanghai Children's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-04
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Severe Sepsis; Sepsis; Septic Shock
Keywords: metabolomics; biomarkers; inflammatory mediator profile; MODS; predictive model
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — 2ml of whole blood collected in sterile tubes containing EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- severe sepsis: patients who diagnosed as sepsis upon PICU admission and develop organ dysfunction during PICU stay
- sepsis: patients recover from sepsis without developing into organ dysfunction

SUMMARY:
In patients diagnosed as sepsis on PICU admission, early and accurate identification of patients who will develop organ dysfunction (severe sepsis) is critical for effective management and positive outcome. A multiple marker approach would improve clinical utility compared with use of a single marker. The primary goal of this part of study is to define a combination of multiple markers, derived from novel biomarkers (nCD-64, IL-27, sTREM, HLA-DR, IL-10), metabolomics and routine clinical parameters, which could predict severe sepsis and determine the severity of disease.

DETAILED DESCRIPTION:
We intend to enroll pediatric sepsis patients at four PICUs and divide them into two groups based on clinical outcomes: severe sepsis group (patients who progress into severe sepsis), sepsis group (patients who do not progress in to severe sepsis). We intend to perform predictive modeling using multivariable analyses of the novel biomarkers and derive a biomarker panel and algorithm for early diagnosis of severe sepsis. The predictive value of the biomarker panel for early identification of severe sepsis will be compared with established indices, such as PRISM III and pSOFA score.

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least two of the following four criteria, one of which must be abnormal temperature or leukocyte count:

  * Coreb temperature of >38.5°C or <36°C.
  * Tachycardia, defined as a mean heart rate >2 SD above normal for age in the absence of external stimulus, chronic drugs, or painful stimuli; or otherwise unexplained persistent elevation over a 0.5- to 4-hr time period OR for children <1 yr old: bradycardia, defined as a mean heart rate <10th percentile for age in the absence of external vagal stimulus, β-blocker drugs, or congenital heart disease; or otherwise unexplained persistent depression over a 0.5-hr time period.
  * Mean respiratory rate >2 SD above normal for age or mechanical ventilation for an acute process not related to underlying neuromuscular disease or the receipt of general anesthesia.
  * Leukocyte count elevated or depressed for age (not secondary to chemotherapy-induced leukopenia) or >10% immature neutrophils
* A suspected or proven (by positive culture, tissue stain, or polymerase chain reaction test) infection caused by any pathogen OR a clinical syndrome associated with a high probability of infection. Evidence of infection includes positive findings on clinical exam, imaging, or laboratory tests

Exclusion Criteria:

* patients without informed consent
* discharge within 48 hours

Ages: 29 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients with sepsis from four tertiary PICUs in Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Severe sepsis | 28 day
  Sepsis plus one of the following: cardiovascular organ dysfunction OR acute respiratory distress syndrome OR two or more other organ dysfunctions
Death | 28 day
  death

SECONDARY OUTCOMES:
secondary infection | 28 day
  infection acquired 48h after PICU admission
length of ICU stay | 28 day
  from PICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, MD, Principal Investigator — Children's Hospital of Fudan University
Locations (4):
- China (4):
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No